CLINICAL TRIAL: NCT05487508
Title: Efficacy of Dexamethasone to Reduce Inflammatory Response and Improve Clinical Outcome in Coronary Artery Bypass Patients: A Multi Arm, Double Blind, Single Center, Randomized Controlled Trial
Brief Title: Efficacy of Dexamethasone to Improve Clinical Outcomes in Coronary Artery Bypass Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dudy Arman Hanafy, Sp. BTKV (K), MARS, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBB.01.01/VII/239/KEP.050/2018
Record Dates: First submitted 2022-07-27; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease; Inflammatory Response
Keywords: dexamethasone; arrhythmia; atrial fibrillation; ventricular tachycardia; ventricular fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac; Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: A double-blind, single center, multi-arm phase 4 randomized controlled clinical trial was conducted with four intervention arms: placebo CCABG, dexamethasone CCABG, placebo OPCAB, and dexamethasone OPCAB arm. The recruitment of subjects were conducted simultaneously by means of a block randomization.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Participants were not aware of the arms/treatment given as they were under general anesthesia during the administration of dexamethasone. Preoperatively, subjects were given explanation of the purpose, methods, benefits, and risks of the procedure including the randomization method. Investigators were kept unaware of the randomization of dexamethasone as they were restricted for assessing the patients' medical record and the patients' identity were coded in the primary database
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexamethasone CCABG (Active Comparator): Dexamethasone administered 1 mg per kg body weight (maximum dose 100 mg), given single dose after induction of anesthesia. Surgeon then carried out the conventional coronary artery bypass graft procedure with the use of cardiopulmonary bypass machine.
  Interventions: Drug: Dexamethasone
- Placebo CCABG (Placebo Comparator): Normal saline (NaCl 0.9%) administered 1 mg per kg body weight (maximum dose 100 mg), given single dose after induction of anesthesia. Surgeon then carried out the conventional coronary artery bypass graft procedure with the use of cardiopulmonary bypass machine.
  Interventions: Drug: Normal saline
- Dexamethasone OPCAB (Active Comparator): Dexamethasone administered 1 mg per kg body weight (maximum dose 100 mg), given single dose after induction of anesthesia. Surgeon then carried out the off-pump coronary artery bypass procedure without the use of cardiopulmonary bypass machine.
  Interventions: Drug: Dexamethasone
- Placebo OPCAB (Placebo Comparator): Normal saline (NaCl 0.9%) administered 1 mg per kg body weight (maximum dose 100 mg), given single dose after induction of anesthesia. Surgeon then carried out the off-pump coronary artery bypass procedure without the use of cardiopulmonary bypass machine.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Administration of intraoperative 1 mg/kg body weight dexamethasone
  Arms: Dexamethasone CCABG; Dexamethasone OPCAB
Drug: Normal saline — Placebo (NaCl 0.9%)
  Arms: Placebo CCABG; Placebo OPCAB

SUMMARY:
This is a single-center, double-blind, randomized controlled clinical trial comparing four groups: placebo conventional coronary artery bypass graft (CCABG) group, dexamethasone CCABG group, placebo off-pump coronary artery bypass (OPCAB) group, and dexamethasone OPCAB group. The primary outcomes of this study is comprised of presence of arrhythmia, major adverse cardiac events (MACE), myocardial infarction, stroke, renal failure, respiratory failure, inflammation, and death. These primary outcomes were assessed during the surgery, 18 hours post surgery, every day during the hospital stay, 14 days and 30 days post surgery.

DETAILED DESCRIPTION:
A single center randomized controlled clinical trial was conducted at Harapan Kita National Cardiovascular Center, Jakarta, Indonesia, as the tertiary cardiovascular referral hospital. The RCT was conducted from July 1st, 2018 to March 31st, 2019 (current status: completed). This study assessed the efficacy of intraoperative high dose dexamethasone administration (1 mg/kg BW, maximum dose 100 mg) in reducing inflammatory response and improving clinical outcome in patients undergoing coronary artery bypass surgery. The study groups consist of placebo CCABG, dexamethasone CCABG, placebo OPCAB, and dexamethasone OPCAB. The subjects were adults indicated to undergo elective coronary artery bypass surgery with no evidence of prior inflammation nor allergic reaction to dexamethasone. Both the patients and the principal investigators were blinded for the treatment-control allocation. The patients were purposively selected and were randomly assigned to one of the arms with block randomization. The primary outcomes of this study is comprised of presence of arrhythmia, major adverse cardiac events (MACE), myocardial infarction, stroke, renal failure, respiratory failure, inflammation, and death. These primary outcomes were assessed during the surgery, 18 hours post surgery, every day during the hospital stay, 14 days and 30 days post surgery. The minimum sample size required for this study was 100 subjects (25 each group).

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease patients indicated for elective coronary artery bypass surgery
* Patients aged >18 years old
* Patients who agreed to participate in this study

Exclusion Criteria:

* Patients with preoperative systemic inflammation evidenced by high axillary temperature (≥38◦C) and high leukocyte count (≥15.000 ul)
* Patients with chronic arrhythmia
* Patients who are indicated to undergo other procedures than coronary artery bypass (i.e. valvular repair, septal repair)
* Patients with history of severe organ dysfunction (class IV congestive heart failure, renal failure, respiratory arrest, and stroke with sequelae)
* Patients with history of cardiac surgery
* Patients who takes routine corticosteroids or immunomodulators
* Patients who are allergic to corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Presence of arrhythmia as seen on EKG | 18 to 24 hours post surgery
  New onset of a postoperative rhythm disorder including atrial fibrillation, ventricular tachycardia, ventricular fibrillation, supraventricular tachycardia, and atrioventricular block
Presence of arrhythmia as seen on EKG | Daily during hospital stay (an average of 7 days)
  New onset of a postoperative rhythm disorder including atrial fibrillation, ventricular tachycardia, ventricular fibrillation, supraventricular tachycardia, and atrioventricular block
Perioperative myocardial infarction as seen on EKG | 18 to 24 hours post surgery
  New Q waves or new left bundle branch block on an electrocardiogram, combined with a biomarker (creatine kinase-MB or troponin) >5 times the upper normal limit
Perioperative myocardial infarction as seen on EKG | Daily during hospital stay (an average of 7 days)
  New Q waves or new left bundle branch block on an electrocardiogram, combined with a biomarker (creatine kinase-MB or troponin) >5 times the upper normal limit
Presence of stroke diagnosed by clinical appearance and CT or MRI | Daily during hospital stay (an average of 7 days)
  A neurologic deficit lasting more than 24 hours with signs of a new ischemic cerebral infarction on computed tomography or magnetic resonance imaging
Renal failure as measured by serum creatinine | 18 to 24 hours post surgery
  Increase in postoperative serum creatinine of at least 3-times the preoperative value, or a serum creatinine level >4mg/dL associated with an acute increase in serum creatinine of at leas 0.5mg/dL

SECONDARY OUTCOMES:
Inflammatory reactions | 18 to 24 hours post surgery
  Measurement of interleukin (IL)-6, C-reactive protein (CRP), and procalcitonin

CONTACTS AND LOCATIONS:
Overall Officials: Komite Etik National Cardiovascular Center Harapan Kita, Study Chair — Ethical Committee of National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, ethical clearance letter, primary database of the study, as well as the study's analysis plan and the manuscript of the study will be made available on the permission by the principal investigator and ethical committee
Supporting Information: Study Protocol, ICF, CSR
Time Frame: September 1st, 2022 for 2 (two) years
Access Criteria: When needed for systematic review or meta analyses of randomized controlled trials

REFERENCES:
- [Background] Dieleman JM, Nierich AP, Rosseel PM, van der Maaten JM, Hofland J, Diephuis JC, Schepp RM, Boer C, Moons KG, van Herwerden LA, Tijssen JG, Numan SC, Kalkman CJ, van Dijk D; Dexamethasone for Cardiac Surgery (DECS) Study Group. Intraoperative high-dose dexamethasone for cardiac surgery: a randomized controlled trial. JAMA. 2012 Nov 7;308(17):1761-7. doi: 10.1001/jama.2012.14144. PMID 23117776